CLINICAL TRIAL: NCT07226154
Title: An Exosomal miRNA Based Predictive Model for Personalized Neoadjuvant Chemotherapy Selection in Pancreatic Ductal Adenocarcinoma
Brief Title: Prediction of Neoadjuvant Chemotherapy Response in Pancreatic Cancer
Acronym: PRECEPT
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19288/PRECEPT
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: PDAC; Exosome; miRNA; FOLFIRINOX; gemcitabine plus nab-paclitaxel; neoadjuvant chemotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Discovery Cohort - NAC Responder Group: Patients with resectable or borderline resectable pancreatic ductal adenocarcinoma (PDAC) who received neoadjuvant chemotherapy (FOLFIRINOX or gemcitabine plus nab-paclitaxel) and achieved a clinical or pathological response.
  Responders were defined as patients showing complete response (CR), partial response (PR), or stable disease (SD) according to radiologic or pathologic assessment after NACT.
  Pre-treatment plasma samples from these patients were analyzed by small RNA sequencing to identify microRNAs associated with favorable chemotherapy response.
  Interventions: Diagnostic Test: Small RNA sequencing
- Discovery Cohort - NAC Non-Responder Group: Patients with resectable or borderline resectable PDAC who received neoadjuvant chemotherapy but demonstrated progressive disease (PD) on radiologic or pathologic evaluation.
  Pre-treatment plasma samples from these patients were analyzed in parallel by small RNA sequencing to identify differential miRNA expression compared with responders.
  Interventions: Diagnostic Test: Small RNA sequencing
- Training Cohort - NAC Responder Group: PDAC patients treated with neoadjuvant chemotherapy (FOLFIRINOX or gemcitabine plus nab-paclitaxel) who achieved CR, PR, or SD responses.
  Candidate microRNAs identified in the Discovery cohort were validated using qRT-PCR (PRECEPT assay).
  Responder group data were used to train and optimize the predictive miRNA panel.
  Interventions: Diagnostic Test: PRECEPT assay (qRT-PCR validation)
- Training Cohort - NAC Non-Responder Group: PDAC patients who received neoadjuvant chemotherapy but exhibited progressive disease (PD).
  Plasma miRNA expression was measured using the PRECEPT assay and compared with responders to refine the predictive model for chemotherapy response.
  Interventions: Diagnostic Test: PRECEPT assay (qRT-PCR validation)
- Validation Cohort - NAC Responder Group: A separate validation cohort of PDAC patients treated with neoadjuvant chemotherapy who achieved CR, PR, or SD.
  The established PRECEPT miRNA panel (qRT-PCR) was applied to evaluate predictive accuracy in this independent responder group.
  Interventions: Diagnostic Test: PRECEPT assay (qRT-PCR validation)
- Validation Cohort - NAC Non-Responder Group: Independent PDAC patients who received neoadjuvant chemotherapy and demonstrated progressive disease (PD).
  This cohort was used to confirm the predictive performance and robustness of the PRECEPT miRNA assay compared with responders.
  Interventions: Diagnostic Test: PRECEPT assay (qRT-PCR validation)

INTERVENTIONS:
Diagnostic Test: Small RNA sequencing — High-throughput small RNA sequencing performed on pre-treatment plasma samples from PDAC patients in the Discovery cohort to identify candidate microRNAs associated with neoadjuvant chemotherapy response. Sequencing data were analyzed to detect differentially expressed miRNAs between responder (CR + PR + SD) and non-responder (PD) groups.
  Groups: Discovery Cohort - NAC Non-Responder Group; Discovery Cohort - NAC Responder Group
Diagnostic Test: PRECEPT assay (qRT-PCR validation) — Quantitative reverse transcription PCR (qRT-PCR)-based validation assay performed on pre-treatment plasma samples in the Training and Validation cohorts. Candidate microRNAs identified in the Discovery cohort by small RNA sequencing were tested using the PRECEPT assay to develop and validate a predictive miRNA panel for neoadjuvant chemotherapy response.
  Groups: Training Cohort - NAC Non-Responder Group; Training Cohort - NAC Responder Group; Validation Cohort - NAC Non-Responder Group; Validation Cohort - NAC Responder Group

SUMMARY:
This study aims to develop and validate a predictive microRNA (miRNA) panel to assess the response to neoadjuvant chemotherapy (NACT) in patients with resectable and borderline resectable pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) remains one of the most lethal malignancies, with a five-year overall survival rate below 12%. Surgical resection combined with systemic chemotherapy offers the best chance for cure; however, only a subset of patients truly benefits from neoadjuvant chemotherapy (NACT). Currently, there are no validated biomarkers to predict response to NACT, making treatment selection largely empirical.

The PRECEPT study (PREdiction of Chemotherapy Effect in Pancreatic Cancer Treatment) aims to identify and validate microRNA (miRNA)-based biomarkers from pre-treatment plasma that can predict therapeutic response to neoadjuvant chemotherapy in patients with resectable or borderline resectable PDAC. Specifically, the study focuses on two standard regimens: FOLFIRINOX and gemcitabine plus nab-paclitaxel (GEM-NABP).

This is a retrospective, non-interventional, observational study using archived plasma samples collected before the initiation of NACT. Exosomal miRNA sequencing (small RNA-seq) has been performed to identify candidate predictive miRNAs. These candidates will be validated using quantitative reverse transcription PCR (qRT-PCR) in an independent patient cohort. The association between miRNA expression levels and pathologic response (CAP grade or tumor regression score) will be analyzed. Additionally, correlations with overall survival (OS) and recurrence-free survival (RFS) will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic ductal adenocarcinoma (PDAC).
* Underwent neoadjuvant chemotherapy (FOLFIRINOX or Gemcitabine/nab-paclitaxel).
* Availability of pre-treatment plasma samples.
* Underwent curative-intent resection (R0 or R1).

Exclusion Criteria:

* Inadequate plasma samples or poor RNA quality for exosomal miRNA analysis.
* Non-adenocarcinoma histology.
* Presence of synchronous or multiple primary malignancies.
* Receipt of chemotherapy regimens other than standard FOLFIRINOX or gemcitabine plus nab-paclitaxel (GEM-NABP).
* Presence of active inflammatory or autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with resectable or borderline resectable pancreatic ductal adenocarcinoma (PDAC) who received neoadjuvant chemotherapy (FOLFIRINOX or Gemcitabine + Nab-paclitaxel) followed by surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Pathological Response Rate | up to 1 year
  Proportion of patients achieving partial or complete pathologic response after neoadjuvant chemotherapy, as assessed using resected pancreatic cancer specimens.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS) | Up to 3 years after surgery
  Time from date of surgical resection to first documented recurrence or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 5 years after surgery
  Time from date of surgical resection to date of death from any cause. Patients alive at last follow-up will be censored.
Radiologic Response Rate | up to 1 year
  Proportion of patients achieving partial or complete radiologic response during neoadjuvant chemotherapy, as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 using contrast-enhanced CT or MRI scans.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Background] Mannucci A, Goel A. Advances in pancreatic cancer early diagnosis, prevention, and treatment: The past, the present, and the future. CA Cancer J Clin. 2026 Jan-Feb;76(1):e70035. doi: 10.3322/caac.70035. Epub 2025 Sep 19. PMID 40971231
- [Background] Hu ZI, O'Reilly EM. Therapeutic developments in pancreatic cancer. Nat Rev Gastroenterol Hepatol. 2024 Jan;21(1):7-24. doi: 10.1038/s41575-023-00840-w. Epub 2023 Oct 5. PMID 37798442
- [Background] Sha M, Gao Y, Yin X, Li X, Liu C, Li S. Engineered exosomes: a promising approach for overcoming challenges in pancreatic cancer therapy. J Nanobiotechnology. 2025 Sep 29;23(1):619. doi: 10.1186/s12951-025-03697-0. PMID 41024179
- [Background] Wang C, Tan G, Zhang J, Fan B, Chen Y, Chen D, Yang L, Chen X, Duan Q, Maimaiti F, Du J, Lin Z, Gu J, Luo H. Neoadjuvant Therapy for Pancreatic Ductal Adenocarcinoma: Where Do We Go? Front Oncol. 2022 Jun 16;12:828223. doi: 10.3389/fonc.2022.828223. eCollection 2022. PMID 35785193
- [Background] Preis M, Gardner TB, Gordon SR, Pipas JM, Mackenzie TA, Klein EE, Longnecker DS, Gutmann EJ, Sempere LF, Korc M. MicroRNA-10b expression correlates with response to neoadjuvant therapy and survival in pancreatic ductal adenocarcinoma. Clin Cancer Res. 2011 Sep 1;17(17):5812-21. doi: 10.1158/1078-0432.CCR-11-0695. Epub 2011 Jun 7. PMID 21652542
- [Background] Philip PA, Lacy J, Portales F, Sobrero A, Pazo-Cid R, Manzano Mozo JL, Kim EJ, Dowden S, Zakari A, Borg C, Terrebonne E, Rivera F, Sastre J, Bathini V, Lopez-Trabada D, Asselah J, Saif MW, Shiansong Li J, Ong TJ, Nydam T, Hammel P. Nab-paclitaxel plus gemcitabine in patients with locally advanced pancreatic cancer (LAPACT): a multicentre, open-label phase 2 study. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):285-294. doi: 10.1016/S2468-1253(19)30327-9. Epub 2020 Jan 14. PMID 31953079
- [Background] Kunzmann V, Siveke JT, Algul H, Goekkurt E, Siegler G, Martens U, Waldschmidt D, Pelzer U, Fuchs M, Kullmann F, Boeck S, Ettrich TJ, Held S, Keller R, Klein I, Germer CT, Stein H, Friess H, Bahra M, Jakobs R, Hartlapp I, Heinemann V; German Pancreatic Cancer Working Group (AIO-PAK) and NEOLAP investigators. Nab-paclitaxel plus gemcitabine versus nab-paclitaxel plus gemcitabine followed by FOLFIRINOX induction chemotherapy in locally advanced pancreatic cancer (NEOLAP-AIO-PAK-0113): a multicentre, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2021 Feb;6(2):128-138. doi: 10.1016/S2468-1253(20)30330-7. Epub 2020 Dec 16. PMID 33338442
- [Background] Labori KJ, Bratlie SO, Andersson B, Angelsen JH, Biorserud C, Bjornsson B, Bringeland EA, Elander N, Garresori H, Gronbech JE, Haux J, Hemmingsson O, Liljefors MG, Myklebust TA, Nymo LS, Peltola K, Pfeiffer P, Sallinen V, Sandstrom P, Sparrelid E, Stenvold H, Soreide K, Tingstedt B, Verbeke C, Ohlund D, Klint L, Dueland S, Lassen K; Nordic Pancreatic Cancer Trial-1 study group. Neoadjuvant FOLFIRINOX versus upfront surgery for resectable pancreatic head cancer (NORPACT-1): a multicentre, randomised, phase 2 trial. Lancet Gastroenterol Hepatol. 2024 Mar;9(3):205-217. doi: 10.1016/S2468-1253(23)00405-3. Epub 2024 Jan 15. PMID 38237621
- [Background] Yeung KTD, Kumar S, Cunningham D, Jiao LR, Bhogal RH. Surgical Outcomes Following Neoadjuvant Treatment for Locally Advanced and Borderline Resectable Pancreatic Ductal Adenocarcinoma. Ann Surg Open. 2024 Sep 4;5(3):e486. doi: 10.1097/AS9.0000000000000486. eCollection 2024 Sep. PMID 39310355
- [Background] Leonhardt CS, Hank T, Pils D, Gustorff C, Sahora K, Schindl M, Verbeke CS, Strobel O, Klaiber U. Prognostic impact of resection margin status on survival after neoadjuvant treatment for pancreatic cancer: systematic review and meta-analysis. Int J Surg. 2024 Jan 1;110(1):453-463. doi: 10.1097/JS9.0000000000000792. PMID 38315795
- [Background] Springfeld C, Ferrone CR, Katz MHG, Philip PA, Hong TS, Hackert T, Buchler MW, Neoptolemos J. Neoadjuvant therapy for pancreatic cancer. Nat Rev Clin Oncol. 2023 May;20(5):318-337. doi: 10.1038/s41571-023-00746-1. Epub 2023 Mar 17. PMID 36932224